CLINICAL TRIAL: NCT00634660
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single, Subcutaneous Doses of rAvPAL-PEG in Subjects With Phenylketonuria
Brief Title: Safety and Tolerability Study of rAvPAL-PEG to Treat Phenylketonuria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAL-001
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 0.001 mg/kg (Active Comparator): One subcutaneous injection of 0.001 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG
- 0.003 mg/kg (Active Comparator): One subcutaneous injection of 0.003 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG
- 0.01 mg/kg (Active Comparator): One subcutaneous injection of 0.01 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG
- 0.03 mg/kg (Active Comparator): One subcutaneous injection of 0.03 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG
- 0.1 mg/kg (Active Comparator): One subcutaneous injection of 0.1 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG
- 0.3 mg/kg (Active Comparator): One subcutaneous injection of 0.3 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG
- 1.0 mg/kg (Active Comparator): One subcutaneous injection of 1.0 mg/kg of rAvPAL-PEG.
  Interventions: Drug: rAvPAL-PEG

INTERVENTIONS:
Drug: rAvPAL-PEG — rAvPAL-PEG will be administered as a single, SC injection at dose levels of 0.001, 0.003, 0.01, 0.03, 0.1, 0.3, and 1.0 mg/kg. The duration of treatment is a single dose of study drug with 42 days (6 weeks) of follow-up.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of injections of rAvPAL-PEG in subjects with PKU.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose study in approximately 35 subjects with PKU who are 16 to 50 years old. Seven cohorts are planned, each consisting of 5 subjects; the cohorts as planned are 0.001, 0.003, 0.01, 0.03, 0.1, 0.3, and 1.0 mg/kg. Increasing doses of rAvPAL-PEG will be assessed sequentially until the final dose is evaluated or any of the stopping criteria are reached. Subjects will each receive a single dose and then will be followed for a total of 42 days (6 weeks) with visits to the clinical research unit (CRU) as specified in the Schedule of Events Toxicity will be measured according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, v 3).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU with both of the following:
* Current blood Phe concentration of ≥600 µmol/L at Screening.
* Average blood Phe concentration of ≥600 µmol/L over the past 3 years, using available data.
* Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
* Willing and able to comply with all study procedures.
* Between the ages of 16 and 50 years, inclusive.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Stable diet with no significant modifications during the 4 weeks preceding the administration of study drug.
* In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Exclusion Criteria:

* Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
* Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
* Any condition that, in the view of the Principal Investigator (PI), places the subject at high risk of poor treatment compliance or of not completing the study.
* Known hypersensitivity to rAvPAL PEG or its excipients.
* Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
* Creatinine above the upper limit of normal.
* Donation of blood or plasma within 30 days prior to the administration of study drug.
* Use of any over-the-counter (OTC) medication, including vitamins, within 7 days prior to the administration of study drug, without evaluation and approval by the Investigator.
* Use of any prescription medication within 14 days prior to the administration of study drug without evaluation and approval by the Investigator.
* Treatment with any drug known to affect hepatic enzyme activity, including (but not limited to) barbiturates, phenothiazines, cimetidine, or carbamazepine, within 30 days prior to study drug administration.
* Use of any tobacco products within 60 days prior to study drug administration.
* Positive urine screen for use of nicotine (cotinine) or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, and opiates).
* Positive test or has been treated for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
• To assess the incidence of treatment-emergent adverse events of a single, subcutaneous (SC) injections of rAvPAL-PEG in subjects with PKU. | 6 weeks
  Specifically, safety was to be assessed by examining the incidence of all treatment-emergent adverse events reported during the study period and clinically significant changes in vital signs and clinical laboratory results, including development of rAvPAL-PEG antibodies.

SECONDARY OUTCOMES:
• To evaluate the pharmacokinetics (PK) of single, SC injections of rAvPAL-PEG administered at escalating doses, in subjects with PKU. | 6 weeks
  Specifically, exposure, AUC- and Cmax -dose proportionality, Tmax , λz and t1/2
• To evaluate the effect of different dose levels of rAvPAL-PEG on blood Phe concentrations in subjects with PKU. | 6 weeks
  Specifically, exposure, AUC- and Cmax -dose proportionality, Tmax , λz and t1/2

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Decker, MD, Study Director — BioMarin Pharmaceutical
Locations (8):
- United States (8):
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Washington University Center for Applied Research Sciences, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No